CLINICAL TRIAL: NCT07276204
Title: A Phase II, Double-masked, Placebo-controlled, Randomized, Parallel Treatment Group Trial to Investigate the Safety and Efficacy of Betaine + Standard of Care (SOC) vs. Placebo + SOC Among Participants With Serologically Diagnosed Metabolic Dysfunction-associated Steatohepatitis (MASH) and Elevated Serum Alanine Aminotransferase (ALT) Level
Brief Title: Betaine vs. Placebo for Serologically Diagnosed Metabolic Dysfunction-associated Steatohepatitis (MASH)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Timothy Morgan, MD, Chief, Hepatology, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Betaine for MASH
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: MASH - Metabolic Dysfunction-Associated Steatohepatitis
Keywords: MASH; ALT; Betaine
MeSH Terms: interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Betaine (Experimental): betaine capsule (oral) 1 gram twice a day
  Interventions: Drug: Betaine
- Placebo (Placebo Comparator): Placebo capsule (oral) twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betaine — Two capsules of betaine, 500 mg, will be consumed twice a day for 24 weeks.
  Arms: Betaine
Drug: Placebo — Two placebo capsules will be taken orally twice a day
  Arms: Placebo

SUMMARY:
The study will evaluate whether betaine reduces liver injury in people with metabolic dysfunction-associated steatohepatitis (MASH). MASH is a type of liver disease that occurs in some people with fatty liver. Betaine is a normal component in the human body and will be taken as a pill.

Seventy (70) participants will be randomized to receive either betaine or placebo for 24 weeks. After stopping treatment, participants will be seen in clinic for another 24 weeks (total participation in the study is approximately 1 year). Procedures performed during the study include blood tests, MRI examinations, questionnaires, and clinic visits.

We will measure improvement in liver injury with blood tests and with MRI.

DETAILED DESCRIPTION:
Study Description: This is a randomized, double-masked phase II trial to test the hypothesis that 24 weeks of treatment with oral betaine, 2 g/day, is a safe and effective treatment for participants with serologically diagnosed metabolic dysfunction-associated steatohepatitis (MASH) and elevated serum alanine aminotransferase (ALT) level.

A total of 70 participants will be randomized at VA Long Beach. Primary endpoint is resolution of at-risk MASH determined by NIS2+™ score at the end of treatment (Week 24). Total study duration for each participant is up to 56 weeks (including screening, treatment, and follow-up).

Primary Objective: To evaluate the efficacy of betaine 2 g/day in reducing liver injury as assessed by percent of participants with NIS2+™ <0.6815 (ie, no longer having at-risk MASH) at the end of treatment (Week 24).

Secondary Objectives:

To evaluate the efficacy of betaine 2 g/day in reducing liver steatosis as assessed by percent of participants with >30% decrease in MRI proton density fat fraction (PDFF) at Week 24 (end of treatment).

To evaluate the safety and tolerability of betaine 2 g/d

Primary Endpoint: The primary endpoint is percent of participants with NIS2+™ <0.6815 (no longer having at-risk MASH) at Week 24 (end of treatment).

Secondary Endpoints:

The percentage of participants with >30% decline in MRI-PDFF at Week 24 (end of treatment).

Safety and tolerability based on adverse events, clinical laboratory values, vital signs, and patient report.

Exploratory Endpoints: There are 5 independent groups of exploratory endpoints: efficacy, cardiovascular risk, laboratory safety, betaine metabolites, and change in behavior and weight.

Study Population: 70 adults of either sex with serologically-diagnosed metabolic dysfunction-associated steatohepatitis and an ALT ≥50 U/L.

Phase: 2 Facilities Enrolling Participants: VA Long Beach Healthcare System Study Intervention: Group 1: betaine (oral, 1 gram BID) + standard of care Group 2: placebo (oral, BID) + standard of care

Study Duration: 5 years

Participant Duration: Participant participation is approximately 13 months:

Treatment: 24 weeks Post-treatment follow-up: 24 weeks

Statistical Assumptions Treatment groups 2 Randomization 1:1 Sample size estimates A two-sided two-sample Z-test with continuity correction and pooled variance Sample size 70 (35 per group) (includes drop outs) Analysis dataset All randomized participants who received at least one does of study medicine

ELIGIBILITY:
Patients must satisfy all the following criteria to be eligible for enrollment.

1. Outpatient
2. Receiving health care at a clinical site that is participating in this trial.
3. A clinical diagnosis of metabolic dysfunction-associated steatotic liver disease based in having 1 or more components of the metabolic syndrome.
4. ALT ≥50 U/L on the most recent measurement and within 28 days prior to randomization
5. NIS2+ ≥0.6815 within 60 days prior to randomization
6. Age 18 to 75 years (inclusive).
7. BMI≥28.
8. MRI PDFF ≥10%.
9. Participants with type 2 diabetes must be receiving stable doses of medicines for the 4 months prior to randomization.
10. Ability to consume oral medication and willing to adhere to the study medicine regimen.
11. Stated willingness to comply with all study procedures, including returning study medicines at each clinic visit, and availability for the duration of the trial.
12. Agreement to adhere to comprehensive lifestyle modification (involving nutrition, exercise, and behavior modification) throughout study duration.
13. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of study medicine administration (ie, after the Week 24 study visit).
14. Provision of a signed and dated informed consent form.

An individual who meets any of the following criteria will be excluded from participating in this trial.

1. Use of FDA-approved medications for the treatment of MASH within the prior 6 months or anticipated to use an FDA-approved medications for MASH during the next 12 months.
2. Use of a glucagon-like peptide-1 receptor agonist (GLP-1 RA) or GLP-1/GIP receptor agonist in the prior 6 months or anticipated use during the next 12 months.
3. Use of a medicine designed to reduce weight within the prior 6 months or anticipated use in the next 12 months.
4. Received insulin within the past 90 days or anticipation of needing insulin in the next 6 months.
5. Uncontrolled diabetes defined as HbA1c of 9.5% or higher within 60 days prior to enrollment.
6. Unstable body weight defined as >5% self-reported (or documented) change in body weight in the period in the 90 days prior to screening.
7. Moderate or heavy alcohol more than 1 week/month during the 3 months prior to screening. Moderate alcohol use is defined as more than 20 g/day (>14 drinks/week) in females or more than 30 g/day (>21 drinks per week) in males. A drink is defined as 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of 80-proof spirits, or the equivalent amount of alcohol in other alcoholic drinks.
8. Phosphatidylethanol (PEth) test > 50 ug/L. (NOTE: PEth will be performed at screening. Participants with PEth >50 ug/L will be excluded. Repeat testing of PEth in participants with a PEth >50 ug/L at screening is not permitted.)
9. Inability to reliably quantify alcohol consumption based upon local study physician judgement.
10. Use of corticosteroids at a does equal to or greater than 10 mg/day of prednisone, for more than 5 days within the prior 30 days.
11. Continued use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks in the 6 months prior to randomization.
12. Cirrhosis of the liver, defined as any of the following:

    * FibroScan® liver stiffness >18 kPa. Note: Participants with FibroScan® liver stiffness between 18 and 20 kPa can be enrolled if they have a liver biopsy that does not demonstrate cirrhosis, provided they do not have another exclusion criteria.
    * MRE liver stiffness >5.0 kPa
    * Prior liver biopsy demonstrating cirrhosis
    * History of esophageal varices, ascites, or hepatic encephalopathy
13. The following laboratory tests during screening (or on blood tests performed within 60 days prior to randomization, if they are not repeated during screening):

    * HDL >46 mg/dL for a male or >58 mg/L for a woman
    * AST or ALT >5 x ULN for the clinical laboratory at the local study site
    * Serum albumin <3.5 g/dL
    * Direct bilirubin >0.6 mg/dL
    * Platelet count less than 125,000 /mm3
    * eGFR < 40 mL/min
    * INR >1.2 (in a participant not receiving anticoagulation medicines)
14. Evidence of other forms of chronic liver disease:

    * Hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg)
    * Hepatitis C as defined by the presence of hepatitis C virus (HCV) RNA or prior treatment for hepatitis C
    * A diagnosis of autoimmune liver disease as defined by compatible liver histology or receipt of treatment for presumed autoimmune liver disease.
    * Primary biliary cholangitis diagnosed by at least 2 of the following Biochemical evidence of cholestasis based mainly on alkaline phosphatase elevation Anti-mitochondrial antibody (AMA) >25 Histological evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts
15. Primary sclerosing cholangitis
16. Known history of Wilson disease, alpha-1-antitrypsin liver disease, or hemochromatosis. Any other type of liver disease that is currently active other than MASH such as drug-induced liver disease, liver cancer, or bile duct obstruction.
17. History of biliary diversion or evidence of current biliary obstruction.
18. Hospitalization for more than 3 days during the prior 60 days.
19. Known positivity for Human Immunodeficiency Virus (HIV) infection.
20. Any of the following in the past: myocardial infarction, stroke, or classification of heart failure New York Heart Association (NYHA) Class II, III, or IV
21. Hospitalization for unstable angina pectoris or transient ischemic attack within 6 months prior to randomization.
22. Current suspected cancer or a prior history of cancer, other than basal cell carcinoma of the skin that was surgically removed.
23. Active, serious medical disease with likely life expectancy less than 5 years
24. Active substance abuse including inhaled or injection drugs in the year prior to screening.
25. Female who is pregnant, breast-feeding, or intends to become pregnant, or is of
26. childbearing potential and not using a highly effective contraceptive method.
27. Current use of choline, betaine, or S-adenosylmethionine supplements, or refusal to abstain from their use during the study.
28. Participation in an IND trial in the 60 days before randomization
29. Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study, including inability to swallow treatment capsules.
30. Failure or inability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
NIS2+ | AT of 24 weeks of treatment with Betaine/Placebo
  The primary endpoint is percent of participants with NIS2+™ <0.6815 (no longer having at-risk MASH) at Week 24 (end of treatment).

SECONDARY OUTCOMES:
MRI-PDFF | at Week 24 (end of treatment).
  The percentage of participants with >30% decline in MRI-PDFF

IPD SHARING:
Plan to Share IPD: No